CLINICAL TRIAL: NCT06675968
Title: A Randomized, Prospective, Single-blind Controlled Clinical Trial to Systematically Assess the Need for Transosseous Anchoring in the Anterolateral Approach to Primary Hip Prosthetic Surgery
Brief Title: Evaluating the Need for Transosseous Anchoring in Anterolateral Hip Prosthetic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mireia Vinas Noguera (Other)
Responsible Party: Sponsor-Investigator, Mireia Vinas Noguera, Doctor, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gluteus Medius
Record Dates: First submitted 2024-10-30; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Suture, Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct suture (Experimental)
  Interventions: Procedure: Direct Suture
- Transsosseus suture (Experimental)
  Interventions: Procedure: Transosseus Suture

INTERVENTIONS:
Procedure: Direct Suture — A capsular closure will be performed, closure of the gluteus medius with a direct tendon and absorbable suture. Addittionally, the iliotibial band, subcutaneous and skin suture closure will be performed.
  Arms: Direct suture
Procedure: Transosseus Suture — A capsular closure will be performed, transosseous suture with a non-absorbable suture. Addittionally, the iliotibial band, subcutaneous and skin suture closure will be performed.
  Arms: Transsosseus suture

SUMMARY:
The study aims to discuss the challenges associated with breakage or failure of the abductor mechanism after total hip arthroplasty, which can lead to gait issues, instability, and the need for revision surgery. Sutures play a crucial role in preventing these failures, with two main types: transosseous and tendon sutures. Transosseous suturing involves using non-absorbable threads anchored in the bone, while tendon suturing uses absorbable threads for layered closure.

Both techniques are commonly used, but there is a lack of evidence to determine which is more beneficial for patients. Current studies are limited and often focus on cases requiring revision surgery due to complications, with transosseous sutures generally being the preferred method.

A meta-analysis indicated that transosseous repair may result in lower dislocation rates and less postoperative pain, but further randomized clinical trials with long-term follow-up are necessary for definitive conclusions. The text proposes a prospective study to compare transosseous suturing with the common absorbable tendon suturing in primary hip surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adult population
* Patients diagnosed with coxarthrosis (stages 2 and 3), confirmed by X-ray, according to D. Tonnis's classification of 1972
* Willingness to follow up for up to 12 months
* Patients capable of understanding the study and giving their informed consent

Exclusion Criteria:

* Difficulty understanding and following the study procedure
* Patients with previous surgery on the same hip
* Patients with a diagnosis other than the inclusion criteria (e.g. acute femoral fracture requiring total hip arthroplasty

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Trendelenburg Test | preoperative and 3 months
  It evaluates the paradoxical elevation of the pelvis in monopodal support on the observed limb. It suggests insufficiency or rupture of the abductor apparatus. It can be positive (+), that is, suggesting abductor pathology, or negative (-), that is, suggesting the absence of a clinical problem in that segment. This is a clinical test that is usually performed during preoperative and follow-up visits to the patient and does not present any risks for the patient. It is performed with the patient standing with body weight evenly distributed. The examiner stands behind the patient and identifies the iliac crests and posterior superior iliac spine. The patient raises the leg that is contralateral to the side being evaluated.

SECONDARY OUTCOMES:
Pain Level | Preoperative at 24 and 48 hours and postoperative at 3, 6 and 12 months
  Pain levels, assessed with a visual analogue scale (VAS) from 0 to 10, with 0 being no pain and 10 being the maximum bearable pain.
Quality of life | Preoperative, 3, 6 and 12 months.
  Functionality and quality of life are assessed with the Harris Hip Score questionnaire (questionnaire on functionality, quality of life, limp, mobility, deformity). This functional test is approved by the International Society of Hip Surgery (Harris Hip Score)
Surgeons sensation | 3 and 12 months
  Score 1-3, 1 suture stability, 2 partial stability, 3 sensation of instability.
Patient Satisfaction | 3 and 12 months
  Questionnaire with 5 possible and gradual responses, from zero to complete satisfaction.
Complications | Up to 1 year
  Determine the presence and, where appropriate, the type.
Complementary tests | Up to 1 year
  In the case of a positive Trendelenburg test, the integrity of the abductor apparatus and motor innervation can be studied. Ultrasound is a non-invasive test usually performed in the case of clinical suspicion of abductor apparatus insufficiency. Electromyography is a non-invasive test, performed using surface electrodes, which assesses the functionality of the superior gluteal nerve, responsible for innervation of the gluteus medius muscle, usually requested in the case of suspicion of the abductor apparatus.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc Taulí, Sabadell, Barcelona, Spain